CLINICAL TRIAL: NCT01653431
Title: Transcranial Direct Current Stimulation to Enhance Cognition in Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Melissa Pigot, Research Assistant, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC12381
Record Dates: First submitted 2012-07-30; First posted 2012-07-31 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Transcranial direct current stimulation (Experimental): Transcranial direct current stimulation combined with cognitive training
  Interventions: Device: Transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator): Sham transcranial direct current stimulation combined with cognitive training
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation

SUMMARY:
The study will examine whether the effects of computerized brain training are enhanced when training is combined with mild brain stimulation in patients with mild cognitive impairment. We hypothesize that this combination will produce greater improvements in cognitive functioning than computerized brain training alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 - 85 years.
* Meet diagnostic criteria for amnestic mild cognitive impairment.

Exclusion Criteria:

* Inability to provide informed consent.
* Concurrent medication likely to affect mental performance.
* Current substance use or dependence in last 3 months.
* Current active psychiatric or neurological condition

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-01; Primary Completion 2018-11 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test II | Post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Martin DM, Mohan A, Alonzo A, Gates N, Gbadeyan O, Meinzer M, Sachdev P, Brodaty H, Loo C. A Pilot Double-Blind Randomized Controlled Trial of Cognitive Training Combined with Transcranial Direct Current Stimulation for Amnestic Mild Cognitive Impairment. J Alzheimers Dis. 2019 Aug 12;71(2):503-512. doi: 10.3233/JAD-190306. PMID 31424410